CLINICAL TRIAL: NCT00667784
Title: Long Term Minor Sibling Donor Well-Being
Status: Terminated | Type: Observational
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0571
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Disorder Related to Bone Marrow Transplantation; Blood Stem Cell Transplant Failure; Disturbance of Emotions Specific to Childhood and Adolescence; Transmission, Blood, Recipient/Donor; Sibling
Keywords: pediatric stem cell donor; emotional sequelae; physical sequelae; psychological consequences of minor donation; Bone Marrow Transplantation; Questionnaire; Survey; Sibling Donor; Stem Cell Transplant; Well-Being
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anxiety Assessment: Minor Donors + Sibling Non-Donors + Parents or Legal Guardians
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires completed before the bone marrow or stem cells are collected, after the transplant, and 6 months after the transplant.
  Other Names: Survey

SUMMARY:
The goal of this research study is to understand what it is like for a young person to have a sick family member and what it is like to donate bone marrow or stem cells for a sick family member.

Primary Aims:

1. Compare minor donor adjustment to minor non-donor adjustment, including anxiety, self-esteem, traumatic stress, achievement, and behavior.
2. Evaluate minor donor adjustment across time, including self -esteem, traumatic stress, anxiety, achievement, and behavior.
3. Investigate the effect of the following on donor well-being:

   * Donor variables: 1) the impact of the harvest, including type of harvest (needle aspiration of bone marrow or peripheral blood stem cell collection by apheresis after injection of G-CSF), pre-procedural anxiety and perceived pain; 2) age of donor at time of transplant, 3) gender, 4) preparedness for transplant, 5) sibling order (for sibling participants), and 6) donor's decision-making and ambivalence regarding donation.
   * Recipient variables: 1) the recipient's level of well-being or death, 2) genetic versus acquired disease types, and 3) familial relationship of donor to recipient.
   * Family support variables: 1) the distress of the family, 2) the quality of the relationship between the potential donor and the recipient, and 3) parent's well-being (post-traumatic stress disorder or PTSD, depression).

Secondary Aim:

Evaluate satisfaction with the donor program.

DETAILED DESCRIPTION:
FOR PARENT or Legal Guardian:

Half of the young persons being asked to participate in this study will be donating bone marrow or stem cells and will be referred to as "minor donors." The other half will not be donating marrow or cells but have a sick family member who will be having a bone marrow or stem cell transplant and will be referred to as "non-donors". For each participating young person, one parent or legal guardian will need to complete the parent questionnaires as well.

You are being asked to participate in this study because you have a sick family member who will have a bone marrow or stem cell transplant at this hospital and you are a caregiver to a healthy child. You will be asked to complete 5 questionnaires shortly before the bone marrow or stem cells are collected, shortly after the transplant, and 6 months after the transplant. You will be asked about your children, family atmosphere, and parental well-being. Most of the questions have a list of possible answers, and you will choose the answer that best describes you. Some questions are left blank for you to write in your answer. It will take about 45 minutes to complete the questionnaires.

FOR CHILD:

If you agree to take part in this study, you will be asked to complete 9 questionnaires shortly before the bone marrow or stem cells are collected, shortly after the transplant, and 6 months after the transplant. You would be asked about your feelings, behavior, and how you are doing in school. These types of questions do not have wrong answers. Most of the questions have a list of possible answers, and you will choose the answer that best describes you. Some questions are left blank for you to write in your answer. It will take about 1 hour to fill out the questionnaires.

Length of Study:

You will participate in the study across a 7 month period. You will begin the study one month before donation and complete the study 6 months after the donation.

This is an investigational study. Up to 30 participants (15 minor donor's parents and 15 non-donor's parents) will be enrolled on this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. sibling of an allogeneic cell therapy transplant patient -- the persons receiving allogeneic transplant may have either an acquired or congenital disease. Acquired diseases include acute lymphoblastic leukemia, acute myelogenous leukemia, severe aplastic anemia, hemoglobinopathies, and lymphomas.Congenital diseases are comprised of hemoglobinopathies and glycogen/lysosomal disorders. Transplant is being considered after failure to respond to traditional therapies or due to the nature of the disease.
2. 5 to 19 years of age
3. speaks English or Spanish
4. one parent or legal guardian willing to participate
5. mentally able to render a valid assessment
6. donor is harvested at this institution
7. donors will participate in the standard psychosocial intervention
8. children in the non-donor group will be matched by age and gender to donor group participants

Exclusion Criteria:

1. participation is limited to one donor per family
2. if a child had matched and declined to donate, that child would not be eligible to participate in the non-donor group

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Parent, legal guardian, or sibling of a patient that will have a bone marrow or stem cell transplant.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Effect of Donor Status on Child's Anxiety (Sibling Donor vs. Sibling Non-Donor) | 7 months (one month pre-donation; one month post-donation; 6 months post-donation)
  Comparison of the two groups (i.e., donor vs. non-donor) using Revised Children's Manifest Anxiety Scale (RCMAS) administered prior to transplant, and two times during course of study to ascertain anxiety. The longitudinal nature of the data necessitates use of a multivariable repeated measures model to examine effects of donor vs. non-donor status on anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Robert, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org